CLINICAL TRIAL: NCT06154629
Title: Effect of a Botanical Ingredient in Healthy Subjects With Anxiety and Poor Sleep Quality
Acronym: Q-Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00034
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-09

CONDITIONS: Poor Quality Sleep
Keywords: botanic extract
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botanical ingredient (Experimental): Consumption for 90 days. Subjects should consume one capsule one hour before going to sleep
  Interventions: Dietary Supplement: Botanical ingredient
- Control Group (Placebo Comparator): Consumption for 90 days. Subjects should consume one capsule one hour before going to sleep
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Botanical ingredient — Consumption for 90 days. Subjects should consume one capsule one hour before going to sleep
  Arms: Botanical ingredient
Dietary Supplement: Control group — Consumption for 90 days. Subjects should consume one capsule one hour before going to sleep
  Arms: Control Group

SUMMARY:
Randomized, controlled, double-blind, single-center clinical trial with two parallel arms depending on the product consumed (experimental product and placebo product) to analyze the efficacy of a botanical extract in reducing anxiety and improving sleep quality.

DETAILED DESCRIPTION:
Subjects who meet the selection criteria will be randomly assigned to each of the study groups (investigational product dose or placebo, depending on the group to which they have been assigned).

The product to be consumed is a botanical extract. Participants will consume the product for 90 days. They should consume one capsule one hour before going to sleep.

They will make a total of five visits to the research laboratory and the tests preestablished in the protocol will be performed. Subsequently, a statistical analysis will be performed with the variables measured in the study to obtain the results.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults.
* Moderate levels of anxiety by STAI.
* Low sleep quality by PSQI.
* Volunteers able to understand the clinical study and willing to comply with its procedures and requirements.

Exclusion Criteria:

* Serious or terminal illness.
* Subjects with body mass index above 32 kg/m2. Pregnant or lactating women.
* Participation in another study involving blood draws or dietary intervention.
* Organic dementias such as Alzheimer's, Huntington's disease, Parkinson's and senile dementia.
* Hypersensitivity to the components of the formula.
* Use of medications that alter cognitive functions or sleep, such as barbiturates, anticonvulsants, benzodiazepines, antidepressants, neuroleptics, alcohol and illicit drugs.
* Subjects with known allergy to some of the study components.
* Inability to understand the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Variation in sleep quality from baseline at 12 weeks. | The evolution of sleep quality after consumption during 12 weeks will be measured.
  Visual analog scale from 0 to 10. The higher the value, the more quality.

SECONDARY OUTCOMES:
Change in Sleep Quality from baseline at 12 weeks | Sleep quality will be measured with a daily scale, from baseline to 12 weeks.
  Visual analog scale from 0 to 10. The higher the value, the more quality.
Sleep quality | It will be measured twice, once at baseline or at the end of the study after 12 weeks of use
  Measured by Pittsburgh test
Sleep efficiency | It will be measured during 4 working days and one weekend day, before starting the consumption of the product and before the end of consumption (90 days).
  Measured by accelerometry, with Actigraph wGT3X-BT
Anxiety questionnaire | Day 1, at 12 weeks later
  Test STAI, to measure the level of anxiety of the subjects
Perceived stress scale | Day 1, at 12 weeks later
  Scale Remor, 2001. Test to measure the level of stress of the subjects
Melatonine | It will be measured twice, once at baseline or at the end of the study after 12 weeks of use
  It is measured with a blood sample in the early evening.
Cortisol | It will be measured twice, once at baseline or at the end of the study after 12 weeks of use
  Measured with blood sample first thing in the morning.
Body composition | The test will be measured at baseline and after 12 weeks of consumption.
  It is a control variable. Measured by bioimpedance
Physical activity control | It will be measured during 4 working days and one weekend day, before starting the consumption of the product and before the end of consumption (90 days).
  It is a control variable. Measured by Actigraph wGT3X-BT
Liver safety variables | It will be measured twice, once at baseline or at the end of the study after 12 weeks.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)
Adverse events | At 12 weeks after consumption
  It will be evaluated at each of the visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain